CLINICAL TRIAL: NCT07008300
Title: Safety, Tolerability, and Pharmacokinetics of an Oral Withania Somnifera Product in Older Adults
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment never started due to time and budgetary constraints
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Alex Speers, ND, Assistant Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00026055; KL2TR002370 (NIH)
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Aging
Keywords: Withania; Herbal Medicine; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told the order in which they receive 120 or 240 mg of the study agent, but every participant will receive 120 mg during the first study period and 240 mg during the second study period. This was done to prevent anticipation of more side effects at the higher dose of the study agent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoden 120 mg (Experimental): Shoden, administered as a single 120 mg capsule, once at the pharmacokinetics visit and once daily for four weeks following the 48 hour visit.
  Interventions: Dietary Supplement: Shoden
- Shoden 240 mg (Experimental): Shoden, administered as a single 240 mg capsule, once at the pharmacokinetics visit and once daily for four weeks following the 48 hour visit.
  Interventions: Dietary Supplement: Shoden

INTERVENTIONS:
Dietary Supplement: Shoden — Shoden® powder is a commercial, dried 70% ethanolic extract of Withania somnifera (ashwagandha, WS) root and leaf, standardized to 35% withanolide glycosides. Shoden® powder is manufactured by Arjuna Natural Pvt Ltd, based in Kochi, Kerala, India.

SUMMARY:
This study will measure the oral bioavailability and pharmacokinetics of known compounds from a standardized Withania somnifera botanical dietary supplement in healthy older adults.

DETAILED DESCRIPTION:
This is a single-blind, crossover trial evaluating (a) the pharmacokinetics of withanolides from two doses (120 and 240 mg) of a commercially available Withania somnifera root and leaf extract (Shoden®), (b) the safety and tolerability of these doses over four weeks' use and (c) the feasibility of remotely measuring sleep- and stress-related outcomes in older adults. There will be two four-week study periods separated by a two-week washout period. During each study period, participants will attend a 13-hour pharmacokinetics study visit, where they will receive a single dose of either 120 or 240 mg Shoden®, and return for 24- and 48-hour blood and urine collections. After the 48-hour visit, they will continue taking Shoden® at the administered dose (120 or 240 mg) for four weeks, at which time they will return for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and older, male and female
2. Body Mass Index (BMI) greater than 17 and less than 35 at screening
3. Sufficient vision and hearing to complete all tests
4. Willingness to discontinue all botanical supplementation for one week prior to and throughout study
5. No known sensitivity to Withania somnifera or any of its derivatives
6. Normal or clinically not significant 12-lead electrocardiogram (ECG) recording
7. Hepatic (ALT, AST, bilirubin), renal (creatinine, estimated GFR), and TSH parameters within normal range
8. Hemoglobin ≥13.0 g/dL or hematocrit ≥39% (males) OR hemoglobin ≥12.5 g/dL or hematocrit ≥38% (females), per FDA recommendations on blood donation
9. General health status that will not interfere with the ability to complete the study
10. Willingness to attend all study visits
11. Willingness to avoid caffeine and xanthine-containing foods or beverages (e.g., coffee, tea, chocolate, caffeine-containing sodas, colas, etc.), as well as grapefruit juice and poppy-containing foods for 48 hours prior to baseline visits
12. Willingness to adhere to special diet (no dairy, grapefruit products, poppy-containing foods, high-fat meals, caffeine, or xanthine-containing foods or beverages) during baseline visits and until after 24-hour visit
13. Mini-Mental State Exam (MMSE) score ≥26

Exclusion Criteria:

1. Current smoking, alcohol, or substance abuse according to DSM-V criteria
2. Participants who are currently pregnant, actively trying to conceive a child, or planning to within three months of study completion
3. Severe aversion to venipuncture
4. Donation of blood within 90 days of screening
5. Participation in drug research study within 90 days of screening
6. Serious health condition (i.e., illness, injury, impairment, or physical or mental condition which requires a) overnight hospitalization or b) continuing treatment that may cause episodic periods of incapacity of more than 3 consecutive days) within 30 days of screening
7. Allergy to nightshade plants (Solanaceae family)
8. Abnormal labs indicating symptomatic and untreated urinary tract infection
9. History of prostate cancer
10. History of kidney transplant
11. Cancer within the last five years, with the exception of non-metastatic skin cancers
12. Comorbid conditions requiring medication such as diabetes, kidney failure, liver failure, hepatitis, blood disorders, hypotension, thyroid disease, respiratory disorders, or cardiovascular disease
13. Presence of sleep apnea, moderate to severe restless leg syndrome, major circadian rhythm changes, or narcolepsy
14. Significant disease of the Central Nervous System (CNS) such as brain tumor, seizure disorder, subdural hematoma, cranial arteritis, or clinically significant stroke
15. Diagnosis of major depression, schizophrenia, bipolar disorder, or other major psychiatric disorder as defined by DSM-V criteria
16. Diseases associated with dementia such as Alzheimer's disease, vascular dementia, normal pressure hydrocephalus or Parkinson's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of withanolides after Shoden administration | For each study period, collected over a 48-hour post-administration period (0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 24 hours, and 48 hours)
  After oral administration of Shoden (120 or 240 mg), plasma concentrations of eleven withanolides (withanolide A, withanolide B, withaferin A, withanone, withanoside IV, withanoside V, 12-deoxywithastramonolide, sominone, viscosalactone B, 4-oxo withaferin A, and 2,3-dihydro-3β-methoxy withaferin-A) will be measured in blood samples obtained over a 48-hour period, using liquid chromatography coupled to multiple reaction monitoring mass spectrometry (LC-MRM-MS) to determine pharmacokinetic parameters (maximum concentration, area under the curve(0-t), and area under the curve(0-infinity)).

SECONDARY OUTCOMES:
Time of maximum concentration of withanolides after Shoden administration | For each study period, collected over a 48-hour post-administration period (0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 24 hours, and 48 hours)
  The time of maximum (tmax) of withanolides will be calculated using liquid chromatography coupled to multiple reaction monitoring mass spectrometry (LC-MRM-MS).
Half-life of withanolides after Shoden administration | For each study period, collected over a 48-hour post-administration period (0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 24 hours, and 48 hours)
  The half-life (t1/2) of withanolides will be calculated using liquid chromatography coupled to multiple reaction monitoring mass spectrometry (LC-MRM-MS).
Steady-state concentration of selected withanolides in plasma | At four weeks for each study period
  Concentration (ng/ml) of selected withanolides in plasma after four weeks' use
Urine concentration of withanolides after Shoden administration | For each study period, collected from 0-12 hours, 24 hours, and 48 hours of each pharmacokinetics visit, and at four weeks
  The concentration (ng/ml) of withanolides in urine will be measured in a pooled urine sample over 12 hours post-Shoden administration, at 24 and 48 hours post-administration, and after four weeks' use.
Adverse events | For each study period, baseline and 12 hours of each pharmacokinetics visit, and at 2 weeks and 4 weeks. Also collected at 2 weeks post-study completion.
  A multi-system questionnaire will record the type and severity (range 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal) of any adverse events. Adverse events will be assessed to determine if any changes are attributable to the study intervention. The proportion of participants who report each type of adverse event will be reported.
Number of participants with abnormal ECG readings | For each study period, baseline (0 hours) and 7 hours of each pharmacokinetics visit, and at 4 weeks.
  Resting electrocardiography will be measured using a ten-lead electrocardiogram. Electrocardiogram changes from the zero-minute (baseline) timepoint will be measured, and alternative clinical explanations considered, in order to determine if any changes are attributable to the study intervention. The investigators will also determine the proportion of all participants who develop changes in electrocardiography compared to the zero-minute timepoint following Shoden administration.
Liver function | For each study period, baseline (0 hours) and at 10 hours of each pharmacokinetics visit, and at 4 weeks
  A comprehensive metabolic panel will measure alanine aminotransferase and aspartate aminotransferase in units per liter as markers of liver function. Enzyme levels falling outside the normal range (0-35 Units per liter for alanine aminotransferase and 17-59 Units per liter for aspartate aminotransferase) will be compared to baseline levels, and alternative clinical explanations considered, in order to determine if elevations are attributable to the study intervention. The investigators will aggregate the measures by using an elevation in either enzyme function as a reflection of overall liver function. The investigators will also determine the proportion of all participants who develop abnormal laboratory values following Shoden administration
Kidney function | For each study period, baseline (0 hours) and at 10 hours of each pharmacokinetics visit, and at 4 weeks
  A comprehensive metabolic panel will measure creatinine and blood urea nitrogen levels in milligrams per deciliter as markers of kidney function. Each parameter falling outside the normal range (0.5 to 1.2 milligrams per deciliter for creatinine and 7 to 20 milligrams per deciliter for blood urea nitrogen) will be compared to baseline values. If elevations are observed, alternative clinical explanations will be considered to determine if elevations are attributable to the study intervention. The investigators will aggregate the measures by using an elevation in either blood urea nitrogen or creatinine as a reflection of overall kidney function. The investigators will also determine the proportion of all participants who develop abnormal laboratory values following Shoden administration
Thyroid-stimulating hormone | For each study period, baseline and at 4 weeks
  Thyroid-stimulating hormone will be measured in units of milli-international units per liter as a marker of thyroid function. Any changes in hormone levels will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in hormone levels are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in thyroid-stimulating hormone following Shoden administration.
Testosterone | For each study period, baseline and at 4 weeks
  Testosterone will be measured in units of nanograms per deciliter. Any changes in hormone levels will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in testosterone levels are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in testosterone following Shoden administration.
White blood cell count | For each study period, baseline and at 4 weeks
  White blood cells will be measured in units of cells per cubic millimeter. Any changes in white blood cell levels will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in white blood cells are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in white blood cells following Shoden administration.
Red blood cell count | For each study period, baseline and at 4 weeks
  Red blood cells will be measured in units of cells per cubic millimeter. Any changes in red blood cell levels will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in red blood cells are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in red blood cells following Shoden administration.
Hemoglobin | For each study period, baseline and at 4 weeks
  Hemoglobin will be measured in grams per deciliter. Any changes in hemoglobin will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in hemoglobin are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in hemoglobin following Shoden administration.
Hematocrit | For each study period, baseline and at 4 weeks
  Hematocrit will be measured in percent. Any changes in hematocrit will be compared to baseline levels. Alternative clinical explanations will be considered in order to determine if any changes in hematocrit are attributable to the study intervention. The investigators will also determine the proportion of all participants who have observed changes in hematocrit following Shoden administration.
Feasibility of administering REDCap surveys | For each study period, baseline and at 4 weeks
  The feasibility of administering REDCap surveys will be assessed by calculating the percentage of administered questionnaires that are returned and fully completed by participants, with feasibility defined as at least 80% of all administered questionnaires returned and completed.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Speers, ND, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual coded participant data that support the published results will be available to be shared for research purposes. Data, plasma, and urine specimens will be stored for future research in a repository. All data/specimens will be coded with each participant's identification code, visit number, and date of collection. Data will be available four months after publication ending five years post article publication.
  For repository requests, the repository guardian Alex Speers (speers@ohsu.edu) or designee will review the requestor's institutional review board approval memo, protocol, and repository sharing agreement before samples/data are released. Separate institutional review board approval/determination will be required for each specific human subject research activity that uses coded data/specimens from the repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available four months after publication, ending five years post-publication.
Access Criteria: For repository requests, the repository guardian will review the requestor's institutional review board approval memo, protocol, and repository sharing agreement before samples/data are released. The Guardian will check for genetic opt out status, withdrawn consent for data/samples, and limitations on future use of data/samples. A signed Repository Sharing Agreement will be collected before data or samples are released. The Repository Guardian will ensure that material transfer agreements for the transfer of biological materials and data use agreements for data shared outside of Oregon Health & Science University are executed as applicable. Specimens and data will be coded with the participant's identification code, visit number, and date of collection. The key for requested specimens and data will be provided separately and with appropriate institutional review board approval.